CLINICAL TRIAL: NCT04774549
Title: Inflammatory Cardiomyopathy Bern Registry
Acronym: FlamBer
Status: Active, not recruiting | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-01100; 2020-01100 (Other: Ethics Comitee)
Record Dates: First submitted 2021-02-18; First posted 2021-03-01 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Myocarditis; Cardiac Sarcoidosis; Pericarditis
Keywords: Myocarditis; Cardiac sarcoidosis; Pericarditis; CMR feature tracking; Strain; T1 and T2 Mapping; LGE; Outcomes; MACE
MeSH Terms: conditions — Myocarditis; Pericarditis; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with inflammatory cardiomyopathy: Patients referred to CMR for suspected/known inflammatory cardiomyopathy and/or diagnosed inflammatory cardiomyopathy from CMR findings

SUMMARY:
Inflammatory cardiomyopathies are associated with inflammation and impaired function of the heart muscle and encompass myo- and pericarditis and cardiac sarcoidosis. Due to the heterogeneity of the clinical manifestations, establishing the diagnosis and prediction of outcome is challenging. Specifically for myocarditis, it is associated with acute and chronic heart failure and sudden cardiac death.

Cardiac magnetic resonance imaging (CMR) allows imaging of tissue characteristics (i.e. edema and fibrosis). CMR is the primary diagnostic tool in myocarditis and can also be used for differentiating other inflammatory diseases. Beside the presence of edema, also hyperemia/capillary leak, fibrosis and myocardial function can be assessed and quantified.

Previous studies demonstrated the prognostic role of CMR features beyond traditional markers of LV function, but are limited to smaller cohorts and single-center studies. Furthermore, CMR is a rapidly developing modality and as new features of the modality become available, additional research is needed to identify which combination of parameters optimize risk stratification of this heterogenous inflammatory cardiomyopathy.

Hence, the goal of the registry is to investigate the diagnostic and prognostic role of clinical techniques in inflammatory cardiomyopathies, particularly CMR, and which combination of features provide the highest potential. This analysis will include new advanced CMR techniques but will also assess the role of other techniques that may be more cost-efficient and more widely available, which could be used as a precursor to CMR imaging exams.

DETAILED DESCRIPTION:
Inflammatory cardiomyopathies, like myocarditis and cardiac sarcoidosis are associated with inflammation of the heart muscle and or pericardium, which is the likely cause of impaired function of the myocardium. Clinical presentation of these diseases present high variability - from asymptomatic cases to patients with cardiac arrest or severe heart failure. Due to the heterogeneity of the clinical manifestations, establishing the diagnosis and prognosis remains challenging.

Due to its high spatial resolution and excellent tissue characterization (i.e. the identification of edema and fibrosis), cardiac magnetic resonance imaging (CMR) is the cornerstone in the workup of acute myocarditis and can also be used for differentiating other inflammatory diseases. One of the main criteria for the non-invasive diagnosis of myocarditis has been the Lake Louise Criteria (LLC), where specifically the inclusion of edema and fibrosis as assessed by CMR are necessary to make the diagnosis of myocarditis. The first recommendations released in 2009 indicated 2 of 3 of the following criteria were needed; presence of edema, hyperemia/capillary leak and/or fibrosis. More recently, 2018 updated guidelines are broadened to non-ischemic inflammation to include sarcoidosis, systemic lupus erythematosus and a variety of types of myocarditis. These criteria now include a 2 of 2 criteria with at least one T2-based (edema) and one T1-based (necrosis/fibrosis mostly) criterion, which can be supported by pericardial effusion or systolic LV wall motion abnormalities.

Further, CMR has been reported to be a very strong prognosticator. Traditional markers such as late gadolinium enhancement (LGE) and left ventricular ejection fraction (LVEF), assessed in CMR are outcome predictors for future adverse cardiac events in myocarditis patients. Similar findings have been shown in sarcoidosis as well. However, CMR is a rapidly developing modality and as new features of the modality frequently become available, additional research is needed to identify the best combination of parameters for risk stratification in patients with inflammatory.

CMR feature tracking (CMR-FT) is a developing contrast-free quantitative method that uses cine images in routinely acquired CMR scanning and it is able to quantify systolic and diastolic myocardial deformation in different orientations. CMR-FT has recently been shown to have diagnostic and prognostic value beyond ejection fraction in patients with coronary artery disease or dilated cardiomyopathy. Recently, the investigators could show in collaboration with the Brigham and Women's Hospital at Harvard Medical School that myocardial strain using CMR-FT provides independent and incremental prognostic value over clinical features, ejection fraction and scar (LGE) in patients with myocarditis. CMR-FT may serve as a novel marker to improve risk stratification in myocarditis. Yet this has not yet been investigated yet with parametric mapping techniques, nor with other inflammatory cardiomyopathies.

The goal of the registry is to investigate the diagnostic and prognostic role of clinical techniques in inflammatory cardiomyopathies, particularly CMR, and which combination of features provide the highest potential. This analysis will include new advanced CMR techniques like feature tracking and T1- and T2 mapping but will also assess the role of other techniques that may be more cost-efficient and more widely available, which could be used as a precursor to CMR imaging exams. Further, other imaging modalities such as echocardiography and nuclear imaging (I.e. Positron Emission Tomography) and computed tomography (CT) findings will be assessed and associated with biomarkers and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Referral to CMR for suspected/known inflammatory cardiomyopathy and/or diagnosed inflammatory cardiomyopathy from CMR findings
* Ability to provide informed consent (knowledge of project languages),
* Age >18 years

Exclusions:

* Inability to give consent or existence of a written or documented oral refusal.
* Evidence of coronary artery disease (CAD) by either previous documented medical history, any imaging findings of CAD, or significant epicardial coronary stenosis by invasive coronary angiography;
* Evidence of hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy, cardiac amyloidosis, Takotsubo cardiomyopathy, Loeffler endocarditis, ventricular noncompaction, cardiac tumor, pulmonary embolism, or persistent severe valve disease.
* Recent cardiovascular surgery or intervention (<90 days prior to CMR)
* Heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to CMR for suspected/known inflammatory cardiomyopathy and/or diagnosed inflammatory cardiomyopathy from CMR findings
Sampling Method: Non-Probability Sample
Enrollment: 1125 (Estimated)
Dates: Start 2005-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
LV (left ventricle) and RV (right ventricle) function as assessed by CMR feature tracking as predictor for MACE (major adverse cardiac Event) | 5 years
  Global and regional longitudinal (%), circumferential (%) and radial (%) strain measurements are used to quantify LV and RV function. MACE is defined as a composite of sustained ventricular tachycardia, recurrent myocarditis, hospitalization for heart failure and all-cause death all-cause death.
LV and RV tissue characterization as assessed by T1 and T2 mapping as predictor for MACE | 5 years
  Global and regional tissue characteristics are assessed by repetitive T1 and T2 mapping (global and regional T1 and T2 time (ms)). MACE is defined as a composite of major cardiovascular endpoints listed above.
Presence of myocardial fibrosis and scar as predictor for MACE | 5 years
  Global and regional myocardial tissue is characterized by gadolinium contrast agent application. The presence and extent (% and total mass (g)) of late gadolinium enhancement is evaluated as a predictor for MACE.

SECONDARY OUTCOMES:
Prognostic impact of sports cessation in acute myocarditis | Repetitive questionnaire at baseline, after 6 and 12 months as well as after 5 years
  Sports behaviour is assessed by repetitive self-evaluating questionnaires before and after diagnosis of acute myocarditis. Sports cessation (total vs. partial vs. no cessation) is evaluated as a predictor of MACE.
Prognostic impact of fragmented QRS in acute myocarditis | 5 years
  Presence and persistence of fragmented QRS as measured by repetitive electrocardiogram is evaluated as a predictor for MACE.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Gräni, MD, PhD, Principal Investigator — Inselspital, Bern University Hospital
Locations (1):
- Department of Cardiology, University Hospital Bern, Inselspital, Bern, Bern, Switzerland

REFERENCES:
- [Background] Grani C, Eichhorn C, Biere L, Murthy VL, Agarwal V, Kaneko K, Cuddy S, Aghayev A, Steigner M, Blankstein R, Jerosch-Herold M, Kwong RY. Prognostic Value of Cardiac Magnetic Resonance Tissue Characterization in Risk Stratifying Patients With Suspected Myocarditis. J Am Coll Cardiol. 2017 Oct 17;70(16):1964-1976. doi: 10.1016/j.jacc.2017.08.050. PMID 29025553
- [Background] Fischer K, Obrist SJ, Erne SA, Stark AW, Marggraf M, Kaneko K, Guensch DP, Huber AT, Greulich S, Aghayev A, Steigner M, Blankstein R, Kwong RY, Grani C. Feature Tracking Myocardial Strain Incrementally Improves Prognostication in Myocarditis Beyond Traditional CMR Imaging Features. JACC Cardiovasc Imaging. 2020 Sep;13(9):1891-1901. doi: 10.1016/j.jcmg.2020.04.025. Epub 2020 Jul 15. PMID 32682718
- [Background] Fischer K, Marggraf M, Stark AW, Kaneko K, Aghayev A, Guensch DP, Huber AT, Steigner M, Blankstein R, Reichlin T, Windecker S, Kwong RY, Grani C. Association of ECG parameters with late gadolinium enhancement and outcome in patients with clinical suspicion of acute or subacute myocarditis referred for CMR imaging. PLoS One. 2020 Jan 10;15(1):e0227134. doi: 10.1371/journal.pone.0227134. eCollection 2020. PMID 31923225
- [Derived] Bernhard B, Tanner G, Garachemani D, Schnyder A, Fischer K, Huber AT, Safarkhanlo Y, Stark AW, Guensch DP, Schutze J, Greulich S, Bastiaansen JAM, Pavlicek-Bahlo M, Benz DC, Kwong RY, Grani C. Predictive value of cardiac magnetic resonance right ventricular longitudinal strain in patients with suspected myocarditis. J Cardiovasc Magn Reson. 2023 Aug 17;25(1):49. doi: 10.1186/s12968-023-00957-6. PMID 37587516
- [Derived] Bernhard B, Schnyder A, Garachemani D, Fischer K, Tanner G, Safarkhanlo Y, Stark AW, Schutze J, Pavlicek-Bahlo M, Greulich S, Johner C, Wahl A, Benz DC, Kwong RY, Grani C. Prognostic Value of Right Ventricular Function in Patients With Suspected Myocarditis Undergoing Cardiac Magnetic Resonance. JACC Cardiovasc Imaging. 2023 Jan;16(1):28-41. doi: 10.1016/j.jcmg.2022.08.011. Epub 2022 Oct 19. PMID 36599567